CLINICAL TRIAL: NCT05200338
Title: Preservation and Transfer of Hepatitis B Virus Immunity After Non-Myeloablative Allogeneic Hematopoietic Stem Cell Transplantation in Adult Sickle Cell Disease Patients (Protect Study)
Brief Title: Preservation and Transfer of HBV Immunity After Allogeneic HSCT for SCD
Acronym: PROTECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Erfan Nur, MD, PhD, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: METC 2021_091
Record Dates: First submitted 2022-01-06; First posted 2022-01-20 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Allogeneic stem cell transplantation; Mixed chimerism; Preservation of immunity; Adoptive transfer of immunity; Hepatitis B virus vaccination
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Engerix-B

STUDY DESIGN:
Intervention Model Description: Prospective observational cohort study. Six SCD patients per cohort will be vaccinated with a recombinant HBV vaccine before allogeneic MSD HSCT (cohort 1a) and haploidentical HSCT (cohort 1b). Six SCD patients not undergoing allogeneic HSCT will be vaccinated as controls (cohort 2). Six haploidentical donors and six matched sibling donors of unvaccinated receivers will be vaccinated against HBV before stem cell donation (cohort 3a and 3b, respectively). All vaccinated patients and the receivers of stem cells of vaccinated donors will receive a booster vaccination at 12 months post-transplantation. Follow-up will be until 2 years post-transplantation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Cohort 1a (Other): SCD patients that are vaccinated against hepatitis B virus before matched sibling donor allogeneic SCT.
  Interventions: Drug: Engerix-B
- Cohort 1b (Other): SCD patients that are vaccinated against hepatitis B virus before haploidentical donor allogeneic SCT.
  Interventions: Drug: Engerix-B
- Cohort 2 (Other): SCD patients that are vaccinated against hepatitis B virus without undergoing allogeneic SCT (control group).
  Interventions: Drug: Engerix-B
- Cohort 3a (Other): SCD patients undergoing matched sibling donor allogeneic SCT whose donor is vaccinated against hepatitis B virus before stem cell collection.
  Interventions: Drug: Engerix-B
- Cohort 3b (Other): SCD patients undergoing haploidentical donor allogeneic SCT whose donor is vaccinated against hepatitis B virus before stem cell collection.
  Interventions: Drug: Engerix-B

INTERVENTIONS:
Drug: Engerix-B — Subjects are vaccinated with an accelerated scheme at 0, +1, +2 months with a booster at +12 months.

SUMMARY:
Sickle cell disease (SCD) patients ending with mixed mononuclear chimerism after non-myeloablative HSCT with alemtuzumab/TBI conditioning will probably preserve their immune response to vaccinations administered prior to the transplantation and will therefore not need to be revaccinated. Furthermore, SCD patients after haploidentical HSCT might benefit from adoptive transfer of immunity from their donors.

To test the first hypothesis, patients undergoing alemtuzumab/TBI HSCT will be vaccinated with a hepatitis B virus (HBV) vaccine before the transplant. To test the second hypothesis, haploidentical and matched related donors will be vaccinated prior to stem cell donation against HBV. Neither the patient nor the donor may previously have been immunized against HBV in all cohorts. Post-transplantation, the investigators will be able to evaluate whether SCD patients preserve their pre-transplant immune response in the post-transplantation period. Furthermore, the investigators will determine whether donors transfer their immunity to HSCT recipients with SCD disease.

DETAILED DESCRIPTION:
Rationale: Sickle cell disease (SCD) is an inherited hemoglobinopathy, characterized by chronic hemolytic anemia and microvascular occlusions leading to pain attacks and progressive deterioration of organ function. As a result, SCD patients have a significantly reduced life expectancy. Allogeneic hematopoietic stem cell transplantation (HSCT) is currently the only available curative treatment for SCD. Recently, a mild non-myeloablative conditioning regimen for HSCT with alemtuzumab (1mg/kg) and low dose (3Gy) total body irradiation (TBI) has been developed for adult SCD patients with a matched sibling donor (MSD) and been implemented in the Netherlands since 2018. The post-transplant setting of SCD patients treated with the alemtuzumab/TBI regimen differs greatly from that in other transplantation regimens usually used as treatment for malignant hematological diseases. Because of its mild character, the conditioning regimen typically results in mixed chimerism. In most patients, stable T-cell donor chimerism of around 50% is achieved. Thus, approximately half of the adaptive immunity is still patient-derived. However, whether these patients preserve their immune response after the transplantation, is not known.

Another promising development is the improvement of HSCT conditioning regimens for adult SCD patients with an haploidentical related donor. At the Amsterdam UMC, haploidentical HSCT has been implemented in 2020 using antithymocyte globulin, fludarabine, cyclophosphamide, thiotepa and low-dose (2Gy) TBI as conditioning regimen and post-transplantation cyclophosphamide (PTCy) as in vivo T-cell depletion. Besides improved engraftment rates, this conditioning regimen is also associated with a reasonably swift immune reconstitution. Unlike the conditioning with alemtuzumab/TBI in MSD HSCT, the above-mentioned conditioning for haploidentical HSCT results in full donor chimerism. Patients losing their immune response due to HSCT might benefit from the transfer of protective immunity from the stem cell donor. Two previous studies have demonstrated the adoption of immunity against hepatitis B virus (HBV) by transplant recipients. However, transplant recipients are also at high risk of gradual disappearance of protective antibodies. In contrast to our study patient population, these studies were conducted in mostly heavily pretreated patients with malignant hematological diseases undergoing myeloablative conditioning regimens.

Currently, it is common practice to revaccinate all patients post-transplant according to the revaccination schedules used for other allogeneic HSCT recipients. However, revaccinating might not be necessary in SCD patients undergoing non-myeloablative HSCT, as they might either preserve their immunity (mixed chimerism after alemtuzumab/TBI conditioning) or benefit from transfer of immunity (haploidentical HSCT)).

The investigators hypothesize, that patients ending with mixed mononuclear chimerism after HSCT will preserve their immune response to vaccinations administered prior to the transplantation and will therefore not need to be revaccinated. Furthermore, the investigators hypothesize, that SCD patients after haploidentical HSCT can benefit from adoptive transfer of immunity from their donors.

To test the first hypothesis, the investigators will vaccinate patients undergoing the alemtuzumab/TBI HSCT with a hepatitis B virus (HBV) vaccine before the transplant. To test the second hypothesis, the investigators will vaccinate haploidentical and matched related donors prior to stem cell donation against HBV. Neither the patient nor the donor may previously have been immunized against HBV in all cohorts. Post-transplantation, the investigators will be able to evaluate whether SCD patients preserve their pre-transplant immune response in the post-transplantation period. Furthermore, the investigators will determine whether donors transfer their immunity to HSCT recipients with SCD disease.

Objectives: Primarily, to investigate whether recipient immunity is preserved and how fast it reconstitutes after non-myeloablative MSD HSCT resulting in mixed chimerism in adult SCD patients. Secondly, to investigate whether donor immunity is transferred to SCD patients after non-myeloablative haploidentical and MSD HSCT.

Study design: Prospective interventional cohort study. Six SCD patients per cohort will be vaccinated with a recombinant HBV vaccine before allogeneic MSD HSCT (cohort 1a) and haploidentical HSCT (cohort 1b). Six SCD patients not undergoing allogeneic HSCT will be vaccinated as controls (cohort 2). Six haploidentical donors and six matched sibling donors of unvaccinated receivers will be vaccinated against HBV before stem cell donation (cohort 3a and 3b, respectively). All vaccinated patients and the receivers of stem cells of vaccinated donors will receive a booster vaccination at 12 months post-transplantation. Follow-up will be until 2 years post-transplantation.

Study population: Adult SCD patients undergoing a matched sibling donor or haploidentical non-myeloablative allogeneic HSCT. HBV naive SCD patients not undergoing HSCT will serve as controls.

Main study parameters/endpoints: Primary endpoint: proportion of SCD patients with a preserved anti-HBs response following non-myeloablative HSCT with an HBV naive MSD. Secondary endpoints: proportion of SCD patients with a preserved HBV specific cellular immune response following non-myeloablative HSCT with an HBV naive MSD. Proportion of SCD patients with a preserved anti-HBs and/or HBV-specific cellular immune response following non-myeloablative HSCT with an haploidentical donor. Proportion of SCD patients adopting their donors anti-HBs and/or HBV-specific cellular immune response following non-myeloablative HSCT. Immune reconstitution as expressed by serum total IgG levels and peripheral blood T-lymphocyte subset counts (CD3+, CD4+, CD8+), B-lymphocyte subset counts (CD19+) and Natural Killer (NK) cell counts at 3-, 6-, 12- and 24-months post-transplantation as compared to baseline (pre-transplantation) values.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* High performance liquid chromatography (HPLC) confirmed diagnosis of SCD (not applicable to participating donors).
* An indication for and a planned matched sibling or haploidentical donor non-myeloablative HSCT at the Amsterdam UMC, location AMC (not applicable to patients in cohort 2 (control group) and participating donors)
* Written informed consent

Exclusion Criteria:

* History of either cleared, chronic or active HBV infection (positive HBsAg, anti-HBs, anti-HBc and/or HBV DNA)
* History of auto-immune diseases and/or use of immunosuppressive drugs
* History of HIV infection
* Known hypersensitivity to yeast of any vaccine constituent
* Donor with a history of HBV infection

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-08 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of SCD patients with a preserved anti-HBs response and HBV-specific cellular response following non-myeloablative allogeneic HSCT with an HBV naive MSD at 12 months post-transplantation as compared to SCD patients without HSCT. | +1 year post-transplantation
  An antibody titer (anti-HBsAg) of >10IU/l is considered protective.

SECONDARY OUTCOMES:
The proportion of SCD patients with a preserved anti-HBs response and HBV-specific cellular response following non-myeloablative allogeneic HSCT with an HBV naive MSD at 3-, 6-, and 24 months post-transplantation as compared to SCD patients without HSCT. | 3-, 6-, and 24 months post-transplantation
The proportion of SCD patients with a preserved anti-HBs response and HBV-specific cellular response following non-myeloablative allogeneic HSCT with an HBV naive haploidentical donor (cohort 1b) at 3-, 6-, 12- and 24 months post-transplantation. | 3-, 6-, 12- and 24 months post-transplantation
The proportion of SCD patients with an adoptive transfer of anti-HBs response and HBV-specific cellular response following non-myeloablative haploidentical HSCT with an HBV vaccinated donor at 3-, 6-, 12- and 24- months post-transplantation (cohort 3a). | 3-, 6-, 12- and 24 months post-transplantation
Serum total IgG level and peripheral blood T-lymphocyte subset counts (CD3+, CD4+, CD8+), B-lymphocyte subset counts (CD19+) and NK cell count, at 3-, 6-, 12- and 24-months post-transplantation as compared to counts before the start of (pre-)conditioning | 3-, 6-, 12- and 24-months post-transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Erfan Nur, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Amsterdam Medical Centre, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided